CLINICAL TRIAL: NCT07155694
Title: Role of Finerenone in African American Veterans With Diabetic Kidney Disease
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Sabyasachi Sen, MD, PhD, Chief of Endocrinology, Washington D.C. Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1780095
Record Dates: First submitted 2025-08-13; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Kidney Disease
Keywords: Empagliflozin; Finerenone; Empagliflozin and Finerenone combination; Podocyte Injury; Chronic Kidney Disease; Diabetic Kidney Disease; Diabetes Mellitus
MeSH Terms: conditions — Diabetic Nephropathies; Renal Insufficiency, Chronic; Diabetes Mellitus | interventions — finerenone; empagliflozin

STUDY DESIGN:
Intervention Model Description: The investigators propose a pilot 2-year, prospective interventional matched open-labeled study enrolling 30 African American veteran patients who come to the DC VAMC nephrology and/or:
  10 subjects will be exposed to Finerenone 10mg orally daily 10 subjects will be exposed to Empagliflozin 10mg orally daily and 10 subjects will be exposed 10mg Finerenone plus 10mg Empagliflozin combination orally daily
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Finerenone (Active Comparator): Finerenone 10mg orally daily for 4 months
  Interventions: Drug: Finerenone 10 MG
- Empagliflozin (Active Comparator): Empagliflozin 10mg orally daily for 4 months
  Interventions: Drug: Empagliflozin 10 MG
- Finerenone and Empagliflozin combination (Active Comparator): Take 10mg Empagliflozin daily, followed by Fineronone 10mg daily after 4 weeks or 1 month of taking empagliflozin. The combination will continue for 3 months or 12 weeks
  Interventions: Drug: Finerenone 10 MG; Drug: Empagliflozin 10 MG

INTERVENTIONS:
Drug: Finerenone 10 MG — Take Finerenone 10 mg orally daily
  Other Names: Kerendia
  Arms: Finerenone; Finerenone and Empagliflozin combination
Drug: Empagliflozin 10 MG — Take Empagliflozin 10 mg orally daily for 4 months
  Other Names: Jardiance
  Arms: Empagliflozin; Finerenone and Empagliflozin combination

SUMMARY:
Primary Objectives: To study podocyte specific injury markers (podocyte specific proteins, PSP) nephrin, podocalyxin and Wilms'Tumor (WT-1) protein in exosomes urine from African American Veterans with albuminuric stage 2 and 3 chronic diabetic kidney disease (DKD), using Empagliflozin or Finerenone or combination therapy.

Secondary Objectives: (1). Correlate changes in exosome-based PSP with standardized biomarkers of kidney injury including urine albumin/creatinine ratio (ACR) and estimated GFR. (2) with systemic inflammatory markers (focusing on vascular and endothelial function) that are already established such as interleukins (IL1, IL6, IL-12), hs-CRP and (3) arterial stiffness measures and with (4) APOL1 mRNA expression levels in peripheral blood derived mononuclear cells (MNC).

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a complex medical condition imposing deleterious effects on multiple organ systems. Prevention of increased cardiovascular mortality and progression to end-stage kidney disease (ESKD) are two major unmet medical needs in patients with CKD, with or without diabetes mellitus, especially in those with albuminuria. In patients with Diabetic Kidney Disease (DKD), the cornerstone of management includes blood pressure control, proteinuria management, maintenance of normal body weight, dietary adherence, and avoidance of nephrotoxic drugs. The management of DKD has undergone extensive changes with the advent of several foundational classes of guideline-based medical therapies (GDMT) for DKD. These include SGLT2i, GLP1-RAs along with Renin-Angiotensin System-inhibitors (RASi). While the benefits of the SGLT2i class of diabetes medications such as Empagliflozin for cardio-kidney outcomes in CKD are well recognized from the landmark EMPA-REG trial, there is less understood in terms of mechanisms of benefit, especially in high-risk patient phenotypes for progression to kidney failure, such as APOL1 positive gene mutation. The results from the recent FIDELIO-DKD and FIGARO-DKD studies showed that finerenone (an aldosterone receptor inhibitor) resulted in a decreased risk of cardiovascular events and slows down CKD progression in patients with type 2 diabetes (T2DM). This was a significant breakthrough and adds an additional class of medication for the treatment of DKD. However, the generalizability of the findings was limited as only 4.7% of the patients were African-American.

The Veterans Health Administration is the largest integrated healthcare system in the USA providing a comprehensive database of patients with CKD. The Nephrology and Endocrinology divisions at DC VAMC manage 175 new CKD patients each month (of whom 70% have diabetes) and 95% are African Americans. African Americans suffer from CKD at significantly higher rates and account for more than 35% of all patients receiving dialysis in the United States. Aggressive management with newer T2DM meds with reno-protective effects is important to be started early. Recently identified genetic variants in the APOL1 gene, found mostly in African Americans may explain a significant proportion of the rising burden of albuminuric CKD in African Americans. APOL1 risk variants G1 and G2 are trypanolytic factors that protect against trypanosomiasis in continental Africa but are associated with a significantly higher risk for the development of podocytopathy and ultimately progressive CKD. Though CKD is quite prevalent in African American patients, the precise mechanism of APOL1 risk variants leading to the progression of DKD in this patient population is unknown and requires further investigation. Interestingly the studies on APOL1 nephropathy have established an association with podocytopathy. Abnormalities in podocyte biology play a central role in the pathogenesis of albuminuric CKD. In CKD with albuminuria, podocyte injury is a key component in the pathophysiology of albuminuric CKD, which is also accompanied by systemic inflammation. The degree of podocyte injury is currently best assessed by kidney biopsy, which is an invasive procedure and not performed in the vast majority of patients with CKD. Therefore, the patterns and extent of podocyte injury in albuminuric CKD is less well understood. The investigators and others have shown improved endothelial function and decreased podocyte-specific urine protein injury markers production with SGLT2i in DKD. Additionally, the literature suggests close crosstalk between the glomerular vascular endothelium and the podocyte. The effect of Finerenone and SGLT2i on markers of podocyte injury, as well as markers of endothelial dysfunction (injury/inflammation) deserve further elucidation, either each medication on its own or in combination in African Americans with proteinuria.

The comparator in this study is Empagliflozin which is a standard of care in DKD. However, the investigators hypothesize that the combination will be more efficacious that either medication alone and synergistic for podocytopathy and proteinuria reversal similar to CONFIDENCE trial even in a CKD prone population of African Americans with diabetes

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of type 2 diabetes (HbA1C at or above 6.5%, or fasting blood glucose of more than 125 or random/ post prandial blood glucose of more than 199mg%)
2. African American veterans
3. Age 20-90 years
4. eGFR ≥25-89 mL/min/1.73 m2 by the CKD-EPI equation)
5. Albuminuria of 30 mg/g or higher
6. BMI=18-39.9
7. Blood pressure controlled to ≤140/90
8. Ability to provide informed consent before any trial related activities are conducted.

Exclusion Criteria

1. If a patient is on statin, need to be on a stable dose for a month.
2. Biopsy proven diagnosis of glomerular disease/glomerulonephritis
3. Active smokers,
4. Active skin wounds undergoing treatment or recent surgery within 1 month (due to possible aberrations in glycemic control)
5. Women who are pregnant, planning to become pregnant, nursing mothers, women of childbearing potential not using birth control measure
6. Hypersensitivity to empagliflozin or finerenone
7. Patients on dialysis
8. eGFR less than 25 mL/min/1.73 m2 by the CKD-EPI equation
9. Planned surgery or planned hospital admission within 5 months of participation in the study
10. At the discretion of PI to ensure health, safety, and well-being of the veteran, participation in this study may be stopped (please see withdrawal criteria)
11. Patients with prior history of diagnosis of heart failure with documented EF of less than 50.
12. Proven diagnosis of Polycystic Kidney Disease.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Urine Exosome Assay | 16 weeks
  To study podocyte specific injury markers (podocyte specific proteins, PSP) nephrin, podocalyxin and Wilms'Tumor (WT-1) protein in exosomes urine on empagliflozin or finerenone or combination therapy. Protein western analysis of Exosomes released from Kidney Podocyte is a indicator of kidney Podocyte health.
  Expressed as a ratio normalized

SECONDARY OUTCOMES:
Renal Function - urine | 16 weeks
  Assessing kidney function by Microalbumin/Creatinine Ratio (Proteinuria) in the urine
Renal Function - serum | 16 weeks
  Estimated glomerular Filtration Rate (Egfr) assessing kidney function based on factors such as creatinine in the serum, age, sex, and ethnicity.
CD34 positive Cell Migratory Function | 16 weeks
  Proportion of cells that migrate through SDF1a in a transwell assay. A larger value indicates better migratory function of the CD34+ cells.
CD34 positive Cell Gene Expression | 16 weeks from visit 1
  Evaluate mRNA gene expression focusing on vascular and endothelial function systemic markers which is normalized to 18s. Fold change of Gene Expression in participants with DKD relative to visit 1.
CD34+ Endothelial Cell Colony Formation Unit (CFU) | 16 weeks
  CFU count of CD34+ endothelial progenitor cells (EPCs)
Arterial Stiffness - Pulse Wave Velocity (PWV) | 16 weeks
  Vessel health assessed by using arterial tonometry with the SphygmoCor CP system from ATCOR.
Arterial Stiffness - Pulse Wave Analysis Augmentation Index | 16 weeks
  Augmentation index was calculated via tonometry with Sphygmocor Device from AtCor (Pulse Wave Analysis). Augmentation index is calculated as the augmentation pressure (the amplitude of the reflected pulse wave) divided by the pulse pressure (systolic - diastolic) * 100 to give a percentage of pulse pressure. The software then calculates an estimated Augmentation Index at heart rate of 75 as a form of "normalization." The higher the values the higher the cardiovascular risk.
Arterial Stiffness - Pulse Wave Analysis Augmentation Pressure | 16 weeks
  Augmentation Pressure is the amplitude of the reflected pulse wave calculated via tonometry with Sphygmocor Device (Pulse Wave Analysis). The higher the values the higher the cardiovascular risk.
Arterial Stiffness - Pulse Wave Analysis Augmentation Index 75 | 16 weeks
  Vessel health is assessed by looking at Arterial stiffness via tonometry. Augmentation index (AI) is defined as the ratio of the augmentation pressure to the pulse pressure, times 100, to give a percentage. Augmentation index 75 normalizes this value to an estimate of the AI at a heart rate of 75bpm. We used Vascular Flow and wave measurement equipment, SphygmoCor Central Pressure system from AtCor. The higher the values the higher the cardiovascular risk.
Hip to Waist Ratio | 16 weeks
  Ratio of Hip to Waist
Body Composition: BMI | 16 weeks
  Body mass index measured using Biometric Impedance Scale in kilogram per square metre
Body Composition: Body Fat Percent | 16 weeks
  Percent of Body Fat measured using Biometric Impedance Tanita Scale
Body Composition: Body Water percent | 16 weeks
  Percent of Body Water measured using Biometric Impedance Tanita Scale
Biochemistry: Hemoglobin A1C (HbA1c) | 16 weeks
  HbA1c percent
Fasting Lipid Profile | 16 weeks
  Measured from a serum blood Lipid Panel: Total Cholesterol, LDL, HDL, and Triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Sabyasachi Sen, MD, PhD, Principal Investigator — Washington DC VA Medical Center
Locations (1):
- Washington DC Veterans Affairs Medical Center (688), Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No